CLINICAL TRIAL: NCT05717413
Title: New Method of Surgical Treatment of Patients With Osteoarthritis of the 1st Metatarsophalangeal Joint
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samara State Medical University (Other)
Collaborators: City Clinical Hospital No.1 named after N.I. Pirogov (Other)
Responsible Party: Sponsor
Other Study IDs: 34
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis
Keywords: modeling of critical loads; geometric model of the foot; Endoprosthesis of 1 metatarsophalangeal joint
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients after arthroplasty of the 1st metatarsophalangeal joint
  Interventions: Device: metatarsophalangeal joint endoprosthesis
- Patients after arthrodesis of the 1st metatarsophalangeal joint

INTERVENTIONS:
Device: metatarsophalangeal joint endoprosthesis — arthroplasty of 1 metatarsophalangeal joint
  Groups: Patients after arthroplasty of the 1st metatarsophalangeal joint

SUMMARY:
Relevance The first metatarsophalangeal joint (MPJ) has an important function in the biomechanics of human gait, especially in the toe and thrust phases, as the full range of motion at this joint provides the body with smooth horizontal acceleration. The flattening of the arches of the foot and, as a result, the overload of its anterior section occupy a leading place in the etiology of deforming osteoarthritis (Hallux rigidus). Hallux rigidus is a disease associated with degenerative changes in the articular cartilage of the first metatarsophalangeal joint. The relevance of the treatment of arthrosis of the first metatarsophalangeal joint is determined by the high incidence and functional significance of the joint.

At the 3rd and 4th degrees of arthrosis, arthrodesis, resection arthroplasty and arthroplasty of the first metatarsophalangeal joint are used.

To date, the most optimal methods of surgical treatment of severe arthrosis of the first metatarsophalangeal joint are arthroplasty and arthrodesis of the joint. These operations are preferred because they achieve good clinical and radiological results. Long-term follow-up studies are needed to confirm the current findings.

Uncoupled endoprostheses are characterized by satisfactory mobility, the ability to withstand high loads, and ligament structures are preserved during their implantation. Of the existing types of non-bonded endoprostheses, zirconium ceramics has a number of advantages, such as: good ingrowth ability, no wear, no rejection reactions. The main advantages of this type of surgical treatment are: rapid pain relief, improved function and stability, individual adaptation of prostheses. Endoprosthetics is recommended for patients of working age with high functional demands.

Thus, the development and implementation of new design solutions in clinical practice is relevant and promising.

task in the surgical treatment of patients with deforming osteoarthritis of the first metatarsophalangeal joint.

Purpose of the study:

To develop and introduce into clinical practice a new method of surgical treatment of patients with deforming osteoarthrosis of the first metatarsophalangeal joint using an anatomically adapted endoprosthesis.

DETAILED DESCRIPTION:
Relevance

The first metatarsophalangeal joint (MPJ) has an important function in the biomechanics of human gait, especially in the toe and thrust phases, as the full range of motion at this joint provides the body with smooth horizontal acceleration. The flattening of the arches of the foot and, as a result, the overload of its anterior section occupy a leading place in the etiology of deforming osteoarthritis (Hallux rigidus). Hallux rigidus is a disease associated with degenerative changes in the articular cartilage of the first metatarsophalangeal joint. The relevance of the treatment of arthrosis of the first metatarsophalangeal joint is determined by the high incidence and functional significance of the joint.

On average, this disease occurs, according to different authors, in 2.5-7.8% of the world population.

Hallux rigidus is a complex disease and numerous conservative and surgical treatments have been developed and described for its treatment. The doctor is faced with the difficult task of choosing an intervention method, for which it is necessary to pay attention to certain criteria: the degree of arthrosis, the age and level of activity of the patient, and the expectation of the result. Conservative treatment can lead to satisfactory performance in selected patients with grade 0 and grade I arthrosis of the first metatarsophalangeal joint with low functional requirements. In the middle stages of arthrosis, an isolated cheilectomy or osteotomy of the proximal phalanx and metatarsal bone is performed, which, despite their differences, for the most part does not lead to a significant increase in the range of motion in the joint. At the 3rd and 4th degrees of arthrosis, arthrodesis, resection arthroplasty and arthroplasty of the first metatarsophalangeal joint are used.

To date, the most optimal methods of surgical treatment of severe arthrosis of the first metatarsophalangeal joint are arthroplasty and arthrodesis of the joint. These operations are preferred because they achieve good clinical and radiological results. Long-term follow-up studies are needed to confirm the current information.

Uncoupled endoprostheses are characterized by satisfactory mobility, the ability to withstand high loads, and ligament structures are preserved during their implantation. Of the existing types of non-bonded endoprostheses, zirconium ceramics has a number of advantages, such as: good ingrowth ability, no wear, no rejection reactions. The main advantages of this type of surgical treatment are: rapid pain relief, improved function and stability, individual adaptation of prostheses. Endoprosthetics is recommended for patients of working age with high functional demands.

Thus, the development and implementation of new design solutions in clinical practice is relevant and promising.

task in the surgical treatment of patients with deforming osteoarthritis of the first metatarsophalangeal joint.

Purpose of the study:

To develop and introduce into clinical practice a new method of surgical treatment of patients with deforming osteoarthrosis of the first metatarsophalangeal joint using an anatomically adapted endoprosthesis.

Research objectives:

1. To evaluate the results of surgical treatment of patients with deforming osteoarthritis of the first metatarsophalangeal joint based on standard approaches.
2. To develop an anatomically adapted all-ceramic endoprosthesis of the first metatarsophalangeal joint.
3. To develop an algorithm for installing a metatarsophalangeal joint endoprosthesis on cadaveric material and the corresponding special tools.
4. Develop specifications for the serial use of the endoprosthesis, including modes of sterilization, packaging and operation.
5. To develop a mode of motor activity in the early postoperative period after the installation of the endoprosthesis of the first metatarsophalangeal joint
6. Conduct a comparative analysis of the mid-term results of the standard and new method of surgical treatment of patients with deforming osteoarthritis of the first metatarsophalangeal joint using the principles of evidence-based medicine.
7. To introduce into clinical practice a new method of surgical treatment of patients with deforming osteoarthrosis of the first metatarsophalangeal joint using anatomically adapted arthroplasty.

Scientific novelty:

For the first time, an anatomically adapted all-ceramic two-component endoprosthesis of the first metatarsophalangeal joint was developed based on the analysis of clinical material and engineering tests.

For the first time, an algorithm for installing an anatomically adapted endoprosthesis of the first metatarsophalangeal joint with the necessary range of surgical special instruments has been developed.

For the first time, a mode of motor activity was developed in the early postoperative period, based on a study of the biomechanics of the first metatarsophalangeal joint after arthroplasty.

For the first time, the advantage of a new method of surgical treatment of patients with arthrosis of the first metatarsophalangeal joint was substantiated using the principles of evidence-based medicine compared to standard methods.

Specifications for the serial use of the endoprosthesis of the first metatarsophalangeal joint in clinical practice have been developed.

A new method of surgical treatment of patients with deforming arthrosis of the first metatarsophalangeal joint has been introduced into clinical practice

Planned scope of research:

1. To assess the mid-term results of surgical treatment of patients with arthrosis of the first metatarsophalangeal joint on the basis of the departments of traumatology and orthopedics of the Clinic of the Samara State Medical University, the trauma department of the State Clinical Hospital No. 1 named after N.I. Pirogov and the Department of Traumatology and Orthopedics of CB "RZD-Medicine".
2. To develop a new anatomically adapted all-ceramic endoprosthesis of the first metatarsophalangeal joint.
3. On the basis of the Samara Regional Bureau of Forensic Medical Examination, develop a method for installing the endoprosthesis of the first metatarsophalangeal joint on cadaveric material.
4. Using a set of studies (clinical, radiological, subometric, plantographic) to give a structural and functional description of the surgical treatment of patients with arthrosis of the first metatarsophalangeal joint in the medium-term postoperative period.
5. To compare the mid-term results of the standard and new method of surgical treatment of patients with deforming osteoarthritis of the first metatarsophalangeal joint using the principles of evidence-based medicine.

Object and methods of research:

The object of the study - patients aged 45 to 70 years. Clinical work will be carried out on the basis of the departments of traumatology and orthopedics of the Clinics of the Samara State Medical University, the trauma department of the State Clinical Hospital No. 1 named after N.I. Pirogov and the Department of Traumatology and Orthopedics of CB "RZD-Medicine". Research work will be carried out using radiation, functional and clinical research methods. It is planned to distribute patients into two groups: control and main. Both groups were comparable in terms of sex, age and duration of the disease. All data will be statistically processed and evaluated from the standpoint of evidence-based medicine. Comparison of functional outcomes will be conducted using the American Association of Foot and Ankle Orthopedics (AOFAS) Clinical Assessment Scale for Foot and Ankle Diseases. A mathematical model and an integral indicator will be built to evaluate the results of surgical treatment.

Expected results:

A new method of surgical treatment of patients with osteoarthritis of the 1st metatarsophalangeal joint will be developed.

A mode of motor activity will be developed in the early postoperative period, based on a study of the biomechanics of the 1st metatarsophalangeal joint after arthroplasty A method for installing an endoprosthesis of the 1st metatarsophalangeal joint will be developed A mathematical model will be built to evaluate the results of treatment of patients with arthrosis of the first metatarsophalangeal joint.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic, post-traumatic and degenerative arthrosis of the first metatarsophalangeal joint
* working age of patients

Exclusion Criteria:

* purulent arthritis and osteomyelitis in the forefoot
* severe osteoporosis
* significant bone defect
* trophic skin changes due to chronic vascular diseases

Ages: 52 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The object of the study - patients aged 45 to 70 years. Clinical work will be carried out in the departments of traumatology and orthopedics of the Clinics of the Samara State Medical University, the trauma department of the State Clinical Hospital No. 1 named after N.I. Pirogov and the Department of Traumatology of CB "RZD-Medicine". Research work includes radiation, functional and clinical research methods. Patients will be divided the control and main groups. Both groups were comparable in terms of sex, age, duration of the disease. All data will be statistically processed according to evidence-based medicine. Comparison of functional outcomes will be conducted using the American Association of Foot and Ankle Orthopedics (AOFAS) Clinical Assessment Scale for Foot and Ankle Diseases.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Dynamics of quality of life indicators using questionnaires | 2 years
  AOFAS scale (American Orthopaedic Foot and Ankle Society Score). The results of treatment are evaluated as follows: excellent - 95-100 points; good - 75-94 points; satisfactory - 51-74 points; bad - 50 points or less.

SECONDARY OUTCOMES:
clinical method | 2 years
  Visual examination, range of motion in the 1st metatarsophalangeal joint, palpation under the heads of the metatarsal bones to identify painful areas
X-ray method | 2 years
  measurement and evaluation of the main x-ray indicators necessary for choosing the method of surgical intervention on the foot, determining the main angles of the foot
Plantography and podometry | 2 years
  determination of the load distribution on the plantar surface of the foot after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinics of Samara State Medical University, Samara, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://samsmu.ru